CLINICAL TRIAL: NCT02000271
Title: Does Vaginal Packing Influence Patient Outcomes Following Vaginal Reconstructive Surgery? A Randomized Controlled Trial
Brief Title: Does Vaginal Packing Influence Patient Outcomes Following Vaginal Reconstructive Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12132-12-089
Record Dates: First submitted 2013-04-30; First posted 2013-12-04 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Vaginal Packing Following Pelvic Reconstructive Surgery

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Vaginal packing (Other): Vaginal packing will be placed as is typical following vaginal reconstructive surgery.
  Interventions: Procedure: Vaginal packing
- No vaginal packing (Experimental): No vaginal packing will be used following vaginal reconstructive surgery.
  Interventions: Procedure: No vaginal packing

INTERVENTIONS:
Procedure: Vaginal packing
  Arms: Vaginal packing
Procedure: No vaginal packing
  Arms: No vaginal packing

SUMMARY:
Vaginal packing is used routinely following vaginal reconstructive surgery. Despite little data to support the practice, purported benefits include reduced pelvic fluid accumulation or blood loss. Patients often complain of discomfort associated with the packing or its removal.

This randomized controlled trial seeks to document differences in subjective impressions of pain in women undergoing vaginal repairs treated with and without packing. The investigators also aim to assess differences in postoperative fluid collection in those with and without packing.

ELIGIBILITY:
Inclusion Criteria:

* Any female aged 18-85 planning to undergo a vaginal hysterectomy with vaginal reconstructive surgery for pelvic organ prolapse, with or without a suburethral sling. Must be able to speak and read English and be able to understand the informed consent.

Exclusion Criteria:

* Undergoing abdominal prolapse repair or repairs not involving hysterectomy, use of mesh, obliterative procedures, concurrent removal of mesh kit, performance of vaginal relaxing incisions, presence of vaginal, uterine, cervical or ovarian malignancy, having a clotting disorder, taking anticoagulation, needing heparin prior to surgery, having intraoperative blood loss greater than 500 cc, or use of regional anesthesia for surgery.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pain and satisfaction | From the first post-operative day up to 6 weeks post-operatively
  Composite of pain and satisfaction as determined by a visual analog scale (validated measure) rating pain as well as a visual analog scale rating satisfaction with either having or not having the vaginal packing placed.

SECONDARY OUTCOMES:
Pelvic fluid collection measurement | In the morning of the first post-operative day.
  Dimensions of pelvic fluid will be measured via transvaginal ultrasound. Length, height, and width will be measured in centimeters
  *This portion of the study has been discontinued due to concerns of patient discomfort during ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- TriHealth Good Samaritan Hospital, Cincinnati, Ohio, United States